CLINICAL TRIAL: NCT03579043
Title: The Effects of Non-Nutritive Sweeteners on Energy Intake
Brief Title: The Effects of Beverages on Food Liking
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment - no eligible participants.
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Major Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: UTK IRB-18-04475-XP
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Coke; Carbonated Water

STUDY DESIGN:
Intervention Model Description: To see if caloric compensation occurs during 3-day exposure to non-nutritive sweeteners, a 3x4 mixed factorial design will be used, with a between-subject factor of intervention group (NNS, NS, and control) and within-subject factor of time (baseline, day 1 of beverage exposure, day 2 of beverage exposure, and day 3 of beverage exposure).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutritive Sweetener (Experimental): Participants will consume 36 ounces of Coke daily for three consecutive days.
  Interventions: Other: Nutritive Sweetener
- Non-Nutritive Sweetener (Experimental): Participants will consume 36 ounces of Diet Coke daily for three consecutive days.
  Interventions: Other: Non-Nutritive Sweetener
- Carbonated Water (Experimental): Participants will consume 36 ounces of carbonated water daily for three consecutive days.
  Interventions: Other: Carbonated Water

INTERVENTIONS:
Other: Nutritive Sweetener — Participants will receive twelve, 12-ounce cans of a beverage that represents their assigned condition. Participants will be instructed to drink their assigned beverages Tuesday through Thursday, and to consume one beverage at 12pm, the second at 3pm, and the third at 6pm. Participants will be instructed that the beverages need to be consumed within +/- 30 minutes of the instructed time. Participants will be instructed that any other beverage consumed on Tuesday through Thursday should be water.
  Other Names: Coke
  Arms: Nutritive Sweetener
Other: Non-Nutritive Sweetener — Participants will receive twelve, 12-ounce cans of a beverage that represents their assigned condition. Participants will be instructed to drink their assigned beverages Tuesday through Thursday, and to consume one beverage at 12pm, the second at 3pm, and the third at 6pm. Participants will be instructed that the beverages need to be consumed within +/- 30 minutes of the instructed time. Participants will be instructed that any other beverage consumed on Tuesday through Thursday should be water.
  Other Names: Diet Coke
  Arms: Non-Nutritive Sweetener
Other: Carbonated Water — Participants will receive twelve, 12-ounce cans of a beverage that represents their assigned condition. Participants will be instructed to drink their assigned beverages Tuesday through Thursday, and to consume one beverage at 12pm, the second at 3pm, and the third at 6pm. Participants will be instructed that the beverages need to be consumed within +/- 30 minutes of the instructed time. Participants will be instructed that any other beverage consumed on Tuesday through Thursday should be water.
  Other Names: Control
  Arms: Carbonated Water

SUMMARY:
The use of non-nutritive sweeteners (NNS) in replacement of nutritive sweeteners (NS) could be a potential weight loss strategy as it may reduce energy intake. One concern with the replacement of NS with NNS is the risk of caloric compensation after consumption of NNS. Most studies have examined the effect of NNS foods and beverages on energy intake in the short-term (one-day or less), with results suggesting lack of compensation in the very short-term (less than one day), and then compensation, or over compensation, when the NNS products are consumed on one day with measures of energy intake taken over 1 to 2 days (Anton et al., 2010; Lavin et al., 1997; Overduin et al., 2016; Appleton et al., 2007; Piernas et al., 2013). Given these mixed results, it is still not clear if NNS foods and beverages are a beneficial strategy for decreasing energy intake. However most studies have been in lab-based settings, in which participants are consuming provided food at specific times. No study has reported on the effect of NNS foods or beverages consumed over several days and energy intake on these days when participants are in free-living situations.

Therefore, the purpose of this investigation is to evaluate how NNS beverage consumption affects energy intake in free-living situations over a span of three days. Through a 3x4 mixed design, participants will be randomized into one of three groups: NNS beverage, NS beverage, or carbonated water (control). Participants will be encouraged to go about their normal daily activities and not change any other aspect except for drink consumption. One baseline and three, 24-hour dietary recalls will be collected over the course of the study to analyze energy intake. The specific aim of this investigation is to determine if caloric compensation occurs during 3-day exposure to NNS beverages.

DETAILED DESCRIPTION:
At the completion of the phone screen, eligible participants will be scheduled to come to the Healthy Eating and Activity Laboratory for the start of their baseline assessment.

The first session will occur the week prior to the test days. At this appointment, informed consent will be obtained, a demographic questionnaire completed, a beverage questionnaire (BEVQ-15) completed, and an appropriate time and preferred mode of contact (text message or e-mail) will be collected. Participant's height and weight will be collected through an electronic scale for weight and a stadiometer for height using standard procedures (Lohman, et al., 1988). Next, participants will be given the SenseWear armband. Participants will be instructed to start wearing the armband upon awakening on Monday morning and to wear the arm band on their upper right arm until going to sleep Monday night (wear time should be at least 10 hours per day). Participants will be instructed to continue wearing the armband, in an identical manner as on Monday, on Tuesday, Wednesday, and Thursday. Participants will be instructed to not alter their physical activity from their normal routine from Monday to Thursday.

Participants will be randomized to one of the three groups, Coke (NS), Diet Coke (NNS), or carbonated water (control) using a random numbers table. For this investigation, Coke and Diet Coke will be used due to Coke and Diet Coke ranked number one and two as the most popular beverages in the U.S. from 2010 to 2018 ("Sweet! America's top 10 brands of soda," 2011; "Top 10 Best Selling Soft Drink Brands in The World," 2016). Next, participants will receive twelve, 12-ounce cans of a beverage that represents their assigned condition. Participants will be instructed to drink their assigned beverages Tuesday through Thursday, and to consume one beverage at 12pm, the second at 3pm, and the third at 6pm. Participants will be instructed that the beverages need to be consumed within +/- 30 minutes of the instructed time. Participants will be instructed that any other beverage consumed on Tuesday through Thursday should be water. Next, instructions will be provided to participants on how to complete the 24-hour dietary recalls and a two-dimensional visual aid will be provided to help participants in estimating portion sizes. Participants will also be given a detailed schedule about their study participation.

Participants will be called on Tuesday, Wednesday, and Thursday to complete 24-hour dietary recalls. Participants will be sent daily reminders regarding their recalls and wearing the armband via text or e-mail (participant preferred mode of contact).

A final appointment will be completed on Friday in the HEAL lab. The armband will be returned and downloaded, the final recall will be completed, and participants will be debriefed about the purpose of the study. Participants will not be responsible for paying for the SenseWear Armband if they lose it or damage it. Once all data are collected, participants will be given a $25 gift card for their participation. If a participant cannot come to the lab on the Friday of their final appointment, then the last recall will be collected via phone and the appointment will be rescheduled in order to collect the armband.

ELIGIBILITY:
Inclusion Criteria:

1. The eligible age range of participants will be 18-35 years. The age range for eligible participants was set because research has shown taste sensitivity declines after the age of 60. In 2001, Mojet and colleagues used sucrose and aspartame to test taste threshold sensitivity in young adults age 19-33 years and elderly adults age 60-75 years. Results showed a decrease in threshold and taste in the elderly adults (Mojet, et al., 2001). Sensitivity to the five basic tastes, sweet, salty, sour, bitter, and umami, begins to decline after the age of 60 ("Aging changes in the senses," n.d.).
2. Individuals with overweight or class I obesity - Body mass index (BMI) range 25-34.9 kg/m2
3. Does not participate in more than 100 minutes of structured, moderate- to high-intensity physical activity weekly
4. Consumes > 36oz of NS beverages daily as assessed by the Beverage Questionnaire (BEVQ)-15 (Hedrick, et al., 2012) - NS beverages include: 100% fruit juice, sweetened juice beverages, energy and sports drinks, sweetened tea or coffee, and soft drinks.
5. Willing to substitute NS beverages for NNS beverages or carbonated water for a three-day period
6. Able to complete all study days consecutively, with all study days following usual schedules and activities (i.e. not traveling)
7. Report a favorable preference for the beverages involved in the study, with participants rating each beverage item ≥3 on a 5-point Likert scale during the phone screen
8. Reports a usual wake up time of 10:00a.m or earlier on Mondays through Fridays.
9. Reports no known allergic reaction to metal

Exclusion Criteria:

1. Report of current dieting or dieting within the past month
2. Report of known reactions to sugar or NNS

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Energy compensation including beverages | 3 test days
  Dietary intake and beverages
Energy compensation not including beverages | 3 test days
  Dietary intake without beverages included

CONTACTS AND LOCATIONS:
Overall Officials: Hannah S Grider, Principal Investigator — University of Tennessee
Locations (1):
- Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anton SD, Martin CK, Han H, Coulon S, Cefalu WT, Geiselman P, Williamson DA. Effects of stevia, aspartame, and sucrose on food intake, satiety, and postprandial glucose and insulin levels. Appetite. 2010 Aug;55(1):37-43. doi: 10.1016/j.appet.2010.03.009. Epub 2010 Mar 18. PMID 20303371
- [Background] Appleton KM, Blundell JE. Habitual high and low consumers of artificially-sweetened beverages: effects of sweet taste and energy on short-term appetite. Physiol Behav. 2007 Oct 22;92(3):479-86. doi: 10.1016/j.physbeh.2007.04.027. Epub 2007 Apr 27. PMID 17540414
- [Background] Hedrick VE, Savla J, Comber DL, Flack KD, Estabrooks PA, Nsiah-Kumi PA, Ortmeier S, Davy BM. Development of a brief questionnaire to assess habitual beverage intake (BEVQ-15): sugar-sweetened beverages and total beverage energy intake. J Acad Nutr Diet. 2012 Jun;112(6):840-9. doi: 10.1016/j.jand.2012.01.023. PMID 22709811
- [Background] Lavin JH, French SJ, Read NW. The effect of sucrose- and aspartame-sweetened drinks on energy intake, hunger and food choice of female, moderately restrained eaters. Int J Obes Relat Metab Disord. 1997 Jan;21(1):37-42. doi: 10.1038/sj.ijo.0800360. PMID 9023599
- [Background] Lohman TR, Roche AF, Martorell R. Anthropometric Standardization Reference Manual. Champaign,Illinois: Human Kinetics Books; 1988.
- [Background] Mojet J, Heidema J, Christ-Hazelhof E. Taste perception with age: generic or specific losses in supra-threshold intensities of five taste qualities? Chem Senses. 2003 Jun;28(5):397-413. doi: 10.1093/chemse/28.5.397. PMID 12826536
- [Background] Overduin J, Collet TH, Medic N, Henning E, Keogh JM, Forsyth F, Stephenson C, Kanning MW, Ruijschop RMAJ, Farooqi IS, van der Klaauw AA. Failure of sucrose replacement with the non-nutritive sweetener erythritol to alter GLP-1 or PYY release or test meal size in lean or obese people. Appetite. 2016 Dec 1;107:596-603. doi: 10.1016/j.appet.2016.09.009. Epub 2016 Sep 9. PMID 27620647
- [Background] Piernas C, Tate DF, Wang X, Popkin BM. Does diet-beverage intake affect dietary consumption patterns? Results from the Choose Healthy Options Consciously Everyday (CHOICE) randomized clinical trial. Am J Clin Nutr. 2013 Mar;97(3):604-11. doi: 10.3945/ajcn.112.048405. Epub 2013 Jan 30. PMID 23364015
- [Background] Sweet! America's top 10 brands of soda. (2011, March 25). Retrieved March 1, 2018, from http://www.nbcnews.com/id/42255151/ns/business-us_business/t/sweet-americas-top-brands-soda/
- [Background] Top 10 Best Selling Soft Drink Brands in The World. (2016, December 30). Retrieved March 1, 2018, from http://www.worldstopmost.com/2017-2018-2019-2020/products/best-selling-soft-drink-brands-world-cheapest-expensive-top-10-popular-list/
- [Background] Aging changes in the senses: MedlinePlus Medical Encyclopedia. (n.d.). Retrieved March 1, 2018, from https://medlineplus.gov/ency/article/004013.htm